CLINICAL TRIAL: NCT03101007
Title: A CLINICAL RANDOMIZED CONTROLLED RSA TRIAL COMPARING THE CEMENTLESS ATTUNE ROTATING PLATFORM KNEE SYSTEM TO THE CEMENTLESS LCS ROTATING PLATFORM KNEE SYSTEM
Brief Title: RSA RCT: Attune RP TKA Versus LCS RP TKA
Acronym: ALKNEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.0027
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis Arthritis; Joint Disease; Musculoskeletal Disease
Keywords: Comparative study; Knee Prosthesis; Prosthesis Design; Treatment Outcome; Follow-up studies; Arthroplast, Replacement, Knee/methods
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ATTUNE (Experimental): Total Knee Replacement Surgery with cementless ATTUNE Rotating Platform Knee Prosthesis by DePuy
  Interventions: Device: ATTUNE Knee Prosthesis by DePuy; Device: LCS Knee Prosthesis by DePuy
- LCS (Active Comparator): Total Knee Replacement Surgery with cementless LCS Rotating Platform Knee Prosthesis by DePuy
  Interventions: Device: ATTUNE Knee Prosthesis by DePuy; Device: LCS Knee Prosthesis by DePuy

INTERVENTIONS:
Device: ATTUNE Knee Prosthesis by DePuy — Total Knee Replacement (TKR) Surgery with cementless ATTUNE rotating platform Knee Prosthesis by DePuy
Device: LCS Knee Prosthesis by DePuy — Total Knee Replacement Surgery with cementless LCS rotating platform Knee Prosthesis by DePuy

SUMMARY:
The LCS Complete Cementless Knee by DePuy Synthes is a rotating platform knee replacement with a good clinical track record and good survival rates.

The cementless ATTUNE Cruciate Sacrificing (CS) Rotating Platform Knee by DePuy Synthes has been designed to provide better range of motion and address the unstable feeling some patients experience during everyday activities, such as stair descent and bending. It is expected that the cementless ATTUNE Rotating Platform Knee will have regulatory approval early 2016. Patient inclusion will start after regular approval has been obtained.

The objective of this study is to accurately assess and compare migration, clinical and radiological outcome and patient reported outcomes (PROMS) of two TKR prostheses: the Cementless ATTUNE Rotating Platform Cruciate Sacrificing Knee System and the LCS Complete Cementless Cruciate Sacrificing Knee System (rotating platform design), both by DePuy Synthes, Warsaw, Indiana, USA. In this single-blind, randomized non-inferiority trial, 32 patients with the ATTUNE Knee System and 32 patients with LCS Knee System will be included.

The study population will consist of patients with symptomatic osteoarthritis of the knee scheduled for TKR surgery at the Department of Orthopaedics, Spaarne Gasthuis, Hoofddorp, The Netherlands. Annually 300 TKA procedures are performed in this department, of which about 95% is Osteo Arthritis (OA). The investigator anticipates that inclusion can be accomplished within a 1 year period and that the total study duration is 3 years.

Main study parameters/endpoints are:

* Migration, measured by means of RSA.
* Patient Reported Outcome Measures by means of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with osteoarthritis and requiring primary knee arthroplasty
* All consecutive patients ("usual care") are included to prevent selection bias in the migration analysis.
* Patient is capable of giving informed consent and expressing a willingness to comply with this study

Exclusion Criteria:

The patient has an a-priori risk for a posterior-stabilized total knee arthroplasty.

* Status after patellectomy
* In case flexion is less than 90 degrees
* The patient is unable or unwilling to sign the Informed Consent specific to this study
* The patient does not understand the Dutch or English language good enough to participate
* Patients indicated for revision arthroplasty
* Patient is diagnosed with rheumatoid arthritis
* When there are not enough markers visible in the baseline RSA photograph and it will not improve by placing the patient in another position, the patient will be excluded from the study (secondary exclusion criteria).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Migration, measured by means of RSA | 2 Years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA).

SECONDARY OUTCOMES:
EQ-5D | 2 Years
  General Health: EuroQol 5 Dimensional (EQ-5D) Health Questionnaire measured using patient questionnaire
KOOS | 2 Years
  Knee Function: Knee injury and Osteoarthritis Outcome Score (KOOS) measured using patient questionnaire
VAS pain | 2 Years
  Pain score after activity and during rest; (Likert scale 0-10)
2 Anchor questions | 2 Years
  Two anchor questions (Likert scale 1-7) about change in functioning and pain since surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rob G Nelissen, Prof PhD MD, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center; Peter A Nolte, PhD MD, Principal Investigator — Dep. Orthopaedics, Spaarne Gasthuis; Edward R Valstar, Prof PhD Msc, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuis, Hoofddorp
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: No